CLINICAL TRIAL: NCT00197028
Title: A Phase I/IIb Randomized, Double-blind, Controlled Study of the Safety, Immunogenicity and Proof-of-concept of RTS,S/AS02D, a Candidate Malaria Vaccine in Infants Living in a Malaria-endemic Region
Brief Title: Examine Safety and Immune Responses of GSK 257049 Vaccine When Administered to Infants Living in a Malaria-endemic Region
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 103967
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2017-04

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine; Engerix-B

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RTS,S/AS02D Group (Experimental): Subjects aged between 6 and 12 weeks at the time of first vaccination received by intramuscular injection a 3-dose vaccination course of RTS,S/AS02D at days 14, 44 and 74 and a 3-dose vaccination course of TETRActHib™ vaccine at days 0, 30 and 60. The RTS,S/AS02D vaccine was administered in the left anterolateral thigh, and the TETRActHib™ vaccine in the right anterolateral thigh.
  Interventions: Biological: RTS,S/AS02D; Biological: TETRActHib™
- Engerix-B Group (Active Comparator): Subjects aged between 6 and 12 weeks at the time of first vaccination received by intramuscular injection a 3-dose vaccination course of Engerix-B® vaccine at days 14, 44 and 74 and a 3-dose of TETRActHib™ vaccine at days 0, 30 and 60. The Engerix-B® vaccine was administered in the left anterolateral thigh, and the TETRActHib™ vaccine in the right anterolateral thigh.
  Interventions: Biological: TETRActHib™; Biological: Engerix-B®

INTERVENTIONS:
Biological: RTS,S/AS02D — 3-dose intramuscular injection in the thigh
  Arms: RTS,S/AS02D Group
Biological: TETRActHib™ — 3-dose intramuscular injection in the thigh.
Biological: Engerix-B® — 3-dose intramuscular injection in the thigh.
  Arms: Engerix-B Group

SUMMARY:
GSK Biologicals is developing in partnership with the Program for Appropriate Technology in Health (PATH) Malaria Vaccine Initiative a candidate malaria vaccine for the routine immunization of infants and children living in malaria endemic areas. The vaccine would offer protection against malaria disease due to the parasite Plasmodium falciparum. The vaccine would also provide protection against infection with hepatitis B virus (HBV).

This trial is being carried out following the demonstration of efficacy of a previous version of the malaria candidate vaccine in children in Mozambique: there, the vaccine demonstrated approximately 30% efficacy against clinical episodes of malaria and approximately 58% efficacy against severe malaria disease.

In order to integrate the malaria vaccine into the Expanded Program on Immunization (EPI) regimen, in malaria-endemic regions, for this trial, a 0.5 ml dose of GSK 257049 vaccine has been developed. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
All infants participating in this phase I/IIb study will receive TETRActHib (a licensed diphtheria-tetanus-pertussis Haemophilus influenzae vaccine manufactured by Aventis Pasteur) by IM injection in their right thigh at 8, 12, and 16 weeks; They will be randomized to receive either the candidate malaria vaccine, GSK 257049 vaccine (0.5 ml dose) or Engerix-B (a licensed hepatitis B vaccine manufactured by GSK Biologicals) by IM injection in their left thigh at 10, 14, 18 weeks. Infants will be followed-up daily for 7 days after each vaccine dose for evaluation of safety and reactogenicity. There will be a 14-day follow-up period after each dose of TETRActHib and after Dose 1 and Dose 2 of GSK 257049 vaccine or Engerix-B, and a one month follow-up period after Dose 3 of GSK 257049 vaccine or Engerix-B for reporting unsolicited symptoms. Serious adverse events will be recorded throughout the 14 month study period. A small amount of blood (2 ml = 1/2 teaspoon) will be obtained at four different time points to measure the immune response elicited by the vaccines administered during this study period. Preliminary indication of vaccine efficacy in this age group will be established by actively monitoring for infection with Plasmodium falciparum.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant of between 6 and 12 weeks of age at the time of first vaccination.
* Written informed consent obtained from the parent(s) or guardian(s) of the subject
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born to a mother who is hepatitis B surface antigen (HBsAg) negative and human immunodeficiency virus (HIV) negative.
* Born after a normal gestation period (between 36 and 42 weeks).
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.

Exclusion Criteria:

* Bacillus Calmette-Guérin tuberculosis vaccine (BCG) administration within one week of proposed administration of a study vaccine.
* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth
* Any chronic drug therapy to be continued during the study period.
* Previous vaccination with diphtheria, tetanus, pertussis, Haemophilus influenzae type b or hepatitis B vaccines.
* Major congenital abnormality.
* Serious acute or chronic illness determined by clinical, physical examination and laboratory screening tests
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of any neurological disorders or seizures.
* Maternal death.
* Hemoglobin < 80 g/L
* Simultaneous participation in any other clinical trial.
* Same sex twin
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trialModerate malnutrition at screening

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2005-08-23; Primary Completion 2007-12-27 (Actual); Study Completion 2007-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Aide P, Aponte JJ, Renom M, Nhampossa T, Sacarlal J, Mandomando I, Bassat Q, Manaca MN, Leach A, Lievens M, Vekemans J, Dubois MC, Loucq C, Ballou WR, Cohen J, Alonso PL. Safety, immunogenicity and duration of protection of the RTS,S/AS02(D) malaria vaccine: one year follow-up of a randomized controlled phase I/IIb trial. PLoS One. 2010 Nov 4;5(11):e13838. doi: 10.1371/journal.pone.0013838. PMID 21079803
- [Background] Aponte JJ, Aide P, Renom M, Mandomando I, Bassat Q, Sacarlal J, Manaca MN, Lafuente S, Barbosa A, Leach A, Lievens M, Vekemans J, Sigauque B, Dubois MC, Demoitie MA, Sillman M, Savarese B, McNeil JG, Macete E, Ballou WR, Cohen J, Alonso PL. Safety of the RTS,S/AS02D candidate malaria vaccine in infants living in a highly endemic area of Mozambique: a double blind randomised controlled phase I/IIb trial. Lancet. 2007 Nov 3;370(9598):1543-51. doi: 10.1016/S0140-6736(07)61542-6. Epub 2007 Oct 18. PMID 17949807
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 103967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103967 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised 2 phases, a double-blind vaccination phase from Month 0 to Month 6, and a single-blind phase (Month 7 to Month 14).
Period: Overall Study
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Started | 107 | 107
Completed | 91 | 86
Not Completed | 16 | 21
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RTS,S/AS02D Group | Engerix-B Group | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.3 (1.42) | 8.3 (1.08) | 8.3 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 59 | 107
  Male | 59 | 48 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs were defined as medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Month 0 to Month 6
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 107 | 107
subjects | 17 | 17

2. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: as for outcome 1
Time Frame: Throughout the entire study period (from Month 0 to Month 14)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 107 | 107
subjects | 35 | 34

3. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HB)
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in milli-international unit per milliliter (mIU/mL). The seroprotection cut-off of the assay was 10 mIU/mL.
Time Frame: Prior to vaccination at Month 0 (PRE) and 1 month post Dose 3 of Engerix-B® or RTS,S/AS02D vaccine (Day 104).
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome variables were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 72 | 70
mIU/mL
  Anti-HB, PRE [N=72;70] | 14.0 [9.6 to 20.5] | 16.6 [11.0 to 25.0]
  Anti-HB, Day 104 [N=68;64] | 10081.6 [7394.9 to 13744.4] | 392.4 [297.0 to 518.5]

4. Secondary Outcome: Concentrations of Anti-circumsporozoite Protein (Anti-CS) Antibodies.
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations are expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The seropositivity cut-off of the assay was 0.5 EL.U/mL.
Time Frame: Prior to vaccination at Month 0 (PRE), 1 month post Dose 3 of Engerix-B® or RTS,S/AS02D vaccine (Day 104) and 3½ months post Dose 3 of Engerix-B® or RTS,S/AS02D vaccine (Day 180).
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 76 | 77
EL.U/mL
  Anti-CS, PRE [N=76;77] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.4]
  Anti-CS, Day 104 [N=71;68] | 199.9 [150.9 to 264.7] | 0.3 [0.2 to 0.3]
  Anti-CS, Day 180 [N=53;61] | 58.8 [41.8 to 82.8] | 0.4 [0.3 to 0.5]

5. Secondary Outcome: Concentrations of Antibodies Against Anti-diphtheria (Anti-D)
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in international unit per milliliter (IU/mL). The seroprotection cut-off of the assay was 0.1 IU/mL.
Time Frame: At Day 90 (1 month post Dose 3 of TETRActHib™ vaccine)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 73 | 72
IU/mL | 1.4 [1.1 to 1.7] | 1.4 [1.2 to 1.7]

6. Secondary Outcome: Concentrations of Antibodies Against Tetanus (Anti-T)
Description: as for outcome 5
Time Frame: At Day 90 (1 month post Dose 3 of TETRActHib™ vaccine)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 73 | 72
IU/mL | 6.2 [5.0 to 7.7] | 5.1 [4.2 to 6.3]

7. Secondary Outcome: Concentrations of Anti-Bordetella Pertussis Toxin Antibodies (Anti-BPT).
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The seropositivity cut-off of the assay was 15 EL.U/mL.
Time Frame: At Day 90 (1 month post Dose 3 of TETRActHib™ vaccine)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 72 | 70
EL.U/mL | 104.4 [89.1 to 122.4] | 106.8 [93.3 to 122.1]

8. Secondary Outcome: Concentrations of Anti-polyribosyl Ribitol Phosphate Antibodies (Anti-PRP).
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per milliliter (µg/mL). The seroprotection cut-off of the assay was 0.15 µg/mL.
Time Frame: At Day 90 (1 month post Dose 3 of TETRActHib™ vaccine)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 73 | 72
µg/mL | 22.1 [16.3 to 29.9] | 17.9 [13.5 to 23.6]

9. Secondary Outcome: Time to First Malaria Infection
Description: Malaria infection by Plasmodium falciparum (P. falciparum) was detected by active detection of infection (ADI) and passive case detection (PCD), and was defined as the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films. The time to first malaria infection is expressed in terms of rate of first malaria infection, that is, the number of malaria infection events reported (n) over the period elapsed until the event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group.
Time Frame: Over the period starting 14 days after Dose 3 of RTS,S/AS02D or Engerix-B® vaccine and extending for 12 weeks thereafter (from Month 2.5 to Month 6)
Population: The analysis was performed on the According-to-Protocol cohort for efficacy, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning efficacy outcome variables were available.
Measure: Number; unit: n/PYAR
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 93 | 92
n/PYAR | 1.01 | 2.67

10. Secondary Outcome: Number of Subjects Prevalent for Plasmodium Falciparum (P. Falciparum)
Description: Subjects prevalent for P. falciparum parasitemia were defined as subjects with the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films.
Time Frame: At Month 6 (3½ months post Dose 3 of RTS,S/AS02D or Engerix-B® vaccine)
Population: as for outcome 9
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 88 | 90
subjects | 4 | 7

11. Secondary Outcome: Plasmodium Falciparum (P. Falciparum) Parasite Density in Subjects Prevalent for Parasitemia
Description: The parasite density in subjects prevalent for P. falciparum parasitemia (subjects with the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films), was detected at a cross sectional time point 3 ½ months after administration of Dose 3 of RTS,S/AS02D or Engerix-B® vaccine (Month 6). Parasite density is expressed as mean, minimum and maximum density in parasite per µL.
Time Frame: At Month 6 (3½ months post Dose 3 of RTS,S/AS02D or Engerix-B® vaccine)
Population: as for outcome 9
Measure: Mean (Full Range); unit: Parasites per µL
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 4 | 7
Parasites per µL | 11573 [131 to 33471] | 10612 [89 to 31993]

12. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain and swelling at injection site.
Time Frame: During the 7 day (Days 0-6) follow-up period after any vaccination with TETRActHib™ vaccine.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available, and whose symptom sheet was completed.
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 107 | 107
subjects
  Pain | 107 | 107
  Swelling | 39 | 47

13. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain and swelling at injection site.
Time Frame: During the 7 day (Days 0-6) follow-up period after any vaccination with Engerix-B® or RTS,S/AS02D vaccine.
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 105 | 106
subjects
  Pain | 105 | 105
  Swelling | 26 | 23

14. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, fever, irritability and loss of appetite. Fever was defined as axillary temperature equal or above (≥) to 37.5 degrees Celsius (C).
Time Frame: During the 7 day (Days 0-6) follow-up period after any vaccination with TETRActHib™ vaccine
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 107 | 107
subjects
  Dorwsiness | 64 | 58
  Fever ≥ 37.5°C | 24 | 25
  Irritability | 89 | 88
  Loss of appetite | 58 | 49

15. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: as for outcome 14
Time Frame: During the 7 day (Days 0-6) follow-up period after any vaccination with Engerix-B® or RTS,S/AS02D vaccine
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 105 | 106
subjects
  Drowsiness | 60 | 69
  Fever ≥ 37.5°C | 25 | 23
  Irritability | 81 | 81
  Loss of appetite | 53 | 62

16. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 14 day (Days 0-13) follow-up period after any vaccination with of TETRActHib™ vaccine
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 107 | 107
subjects | 64 | 51

17. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: as for outcome 16
Time Frame: During the 14 day (Days 0-13) follow-up period after vaccination with any among Doses 1 and 2 of Engerix-B® or RTS,S/AS02D vaccine.
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 105 | 106
subjects | 50 | 47

18. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: as for outcome 16
Time Frame: During the 30 day (Days 0-29) follow-up period after vaccination with Dose 3 of Engerix-B® or RTS,S/AS02D vaccine.
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Number analyzed (Participants) | 97 | 97
subjects | 32 | 39

ADVERSE EVENTS:
Time Frame: SAEs: entire study period (Months 0-14); Unsolicited AEs: Days 0-13 or 0-29 periods (as specified in notes); Solicited local/general symptoms: 7 day (Days 0-6) follow-up period after any vaccination.
Description: For solicited symptoms and unsolicited AEs assessed following vaccination, the number of participants at risk included those vaccinated subjects from the Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | RTS,S/AS02D Group | Engerix-B Group
Serious Adverse Events (participants affected / at risk) | 35/107 | 34/107
Other Adverse Events (participants affected / at risk) | 107/107 | 107/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTS,S/AS02D Group (N=107) | Engerix-B Group (N=107)
Gastroenteritis (Infections and infestations) | 13 | 18
Anaemia (Blood and lymphatic system disorders) | 17 | 13
Plasmodium falciparum infection (Infections and infestations) | 15 | 13
Bronchopneumonia (Infections and infestations) | 4 | 5
Bronchitis (Infections and infestations) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Pneumonia (Infections and infestations) | 4 | 3
Marasmus (Metabolism and nutrition disorders) | 2 | 2
Oral candidiasis (Infections and infestations) | 2 | 1
Otitis media (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Febrile convulsion (Nervous system disorders) | 1 | 1
Pyoderma (Infections and infestations) | 1 | 2
Pyrexia (General disorders) | 0 | 2
Ascariasis (Infections and infestations) | 0 | 1
Bronchial hyper reactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Tinea capitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | RTS,S/AS02D Group (N=107) | Engerix-B Group (N=107)
Pain (General disorders) | 107 | 107 — During the 7-day follow-up period after vaccination with TETRAct/Hib vaccine
Swelling (General disorders) | 39 | 47 — During the 7-day follow-up period after vaccination with TETRAct/Hib vaccine
Drowsiness (General disorders) | 64 | 58 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Fever (General disorders) | 24 | 25 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Irritability (General disorders) | 89 | 88 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Loss of appetite (General disorders) | 58 | 49 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Upper respiratory tract infection (Infections and infestations) | 26 | 18 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 10 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Malaria (Infections and infestations) | 14 | 7 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Bronchitis (Infections and infestations) | 7 | 5 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Anaemia (Blood and lymphatic system disorders) | 11 | 4 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Conjunctivitis (Eye disorders) | 7 | 2 — During the 14-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Diarrhea (Gastrointestinal disorders) | 17 | 6 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine
Upper respiratory tract infection (Infections and infestations) | 21/105 | 24/106 — During the 14-day follow-up period after vaccination with Doses 1 and 2 of RTS,S/AS02D or Engerix-BTM vaccine
Upper respiratory tract infection (Infections and infestations) | 7/97 | 15/97 — During the 29-day follow-up period after vaccination with Dose 3 of RTS,S/AS02D or Engerix-BTM vaccine
Malaria (Infections and infestations) | 3/105 | 7/106 — During the 14-day follow-up period after vaccination with Doses 1 and 2 of RTS,S/AS02D or Engerix-B® vaccine
Pyrexia (General disorders) | 5/97 | 3/97 — During the 29-day follow-up period after vaccination with Dose 3 of RTS,S/AS02D or Engerix-B® vaccine
Diarrhea (Gastrointestinal disorders) | 8/105 | 8/106 — During the 14-day follow-up period after vaccination with Doses 1 and 2 of RTS,S/AS02D or Engerix-B® vaccine
Diarrhea (Gastrointestinal disorders) | 6/97 | 6/97 — During the 29-day follow-up period after vaccination with Dose 3 of RTS,S/AS02D or Engerix-B® vaccine
Pain (General disorders) | 105/105 | 105/106 — During the 7-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Swelling (General disorders) | 26/105 | 23/106 — During the 7-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Drowsiness (General disorders) | 60/105 | 69/106 — During the 7-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Fever (General disorders) | 25/105 | 23/106 — During the 7-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Irritability (General disorders) | 81/105 | 81/106 — During the 7-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Loss of appetite (General disorders) | 53/105 | 62/106 — During the 7-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Malaria (Infections and infestations) | 0/97 | 7/97 — During the 30-day follow-up period after vaccination with RTS,S/AS02D or Engerix-B® vaccine
Ear infection (Infections and infestations) | 3 | 6 — During the 14-day follow-up period after vaccination with TETRAct/Hib vaccine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.